CLINICAL TRIAL: NCT06154681
Title: Effectiveness of a World Digital Detox Program for Enhancing Youth and Family Well-being: A Multicenter Randomized Controlled Trial
Brief Title: World Digital Detox Program for Enhancing Youth and Family Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innowage Limited (Industry)
Collaborators: Zep Foundation (Unknown); Aarogyam UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Zep-WDDD-I 01
Record Dates: First submitted 2023-11-16; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Psychological Well-Being; Adolescent Behavior; Family
MeSH Terms: conditions — Psychological Well-Being; Adolescent Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- World Digital Detox Family Program (Experimental): The 4-week Self-Help World Digital Detox Family and Society Program is a comprehensive program, with variety of self-guided activities, discussions, and reflection exercises. The intervention encompasses both individual and collective components.
  Interventions: Other: World Digital Detox Family Program
- Wait-list Control (No Intervention): Wait-list control group underwent the standard assessment and screening process but not engaged in the intervention during the 4-week period.

INTERVENTIONS:
Other: World Digital Detox Family Program — The Self-Help World Digital Detox Family Program spans four weeks and offers a structured approach to tackle the rising issues associated with the overuse of screens, social media, and digital devices within families. This intervention provides practical tools and strategies to be implemented on a weekly basis.
  Arms: World Digital Detox Family Program

SUMMARY:
The pervasive presence of digital devices and technology has reshaped contemporary society, providing numerous benefits but also prompting concerns about prolonged screen time, particularly with smartphones and social media. These concerns extend to their impact on interpersonal relationships and mental well-being. The Zep Foundation's World Digital Detox Program to address the challenges posed by excessive screen exposure, social media usage, and digital screen dependency.

This study aimed to assess the efficacy of the digital detox family intervention, endorsed by the World Digital Detox Day program, in curbing the use of digital devices-specifically smartphones and social media-and enhancing the overall well-being of youth and families.

ELIGIBILITY:
Inclusion Criteria:

for Caregivers:

* Age 18 or older at baseline assessment;
* Primary caregiver responsible for the care of an adolescent 10-14 who is a resident in the same household
* Able to speak English
* Agreement to participate in the program;
* Consent for self and child to participate in the study.

for Adolescents:

* Age 10-14 at baseline assessment;
* Agreed to participate in the study;
* Caregiver consent to participate in the study.

Exclusion Criteria:

* Serious Medical Conditions requiring frequent hospitalization
* Special Educational Need Children and Adolescents
* Substance abuse

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) | From baseline to 4-week post intervention
  The 10-item PSS was used to assess perception of stress.

SECONDARY OUTCOMES:
Media Multitasking-Revised (MMT-R) scale | From baseline to 4-week post intervention
  18-item MMT-R scale measured proactive behaviors of compulsive or inappropriate phone use as well as more passive behaviors
Family Communication Scale (FCS) | From baseline to 4-week post intervention
  10-item FCS was used to measure satisfaction toward the aspects of positive communication among family members
Family Health Behaviours Scale (FHBS) | From baseline to 4-week post intervention
  27-items FHBS scale includes the subscales to assess parental behavior, meal routines, physical activity, and children's behavior.
Mental Health Continuum Short Form (MHC-SF) | From baseline to 4-week post intervention
  14-items MHC-SF measure the adult's emotional, psychological, and social well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Rekha Chaudhari, PhD, Study Director — World Digital Detox Day, Zep Foundation; Neha Sharma, PhD, Study Chair — Aarogyam UK
Locations (1):
- World Digital Detox Day, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided